CLINICAL TRIAL: NCT05416619
Title: Effects of Hand MOtor Rehabilitation Using a sEMG-biofeedback, After Stroke: a Longitudinal Pilot Study
Brief Title: Effects of Hand MOtor Rehabilitation Using a sEMG-biofeedback
Acronym: MORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Andrea Turolla, Principal Investigator, IRCCS San Camillo, Venezia, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016.29.1
Record Dates: First submitted 2022-05-31; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic; Hemiparesis
Keywords: Neurological Rehabilitation; Hand Recovery; Electromyography
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: Intervention is provided by a wearable device for hand rehabilitation. The device is composed by 8 bipolar electrodes that are able to detect muscle activation to control a computer interface to execute sEMG-biofeedback training for hand motor recovery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sEMG-biofeedback Group (Experimental): Receive 1 hour of sEMG-biofeedback hand training provided by wearable REMO® and 1 hour of daily conventional rehabilitation therapy.
  Interventions: Device: REMO®

INTERVENTIONS:
Device: REMO® — The patients receive daily 1 hour of conventional therapy and 1 hour of treatment of REMO®, that is a wearable composed by 8 bipolar electrodes able to detect the surface electromyography of the forearm muscles. REMO® allows the control of a computer interface using the surface electromyography to execute sEMG-biofeedback exercises for hand rehabilitation. The movements required for hand rehabilitation are the following: thumb abduction, pinch, finger flexion, finger extension, wrist flexion, wrist extension, forearm pronation, forearm supination, radial wrist deviation and ulnar wrist deviation. The treatment consists in 15 sessions, 1hour/day, for 5 days/week, for 3 weeks. The patients are clinically evaluated before and after the REMO® treatment.

SUMMARY:
Stroke is the first cause of disability worldwide. The motor impairment of the hand is one of the most common sequelae in patients after stroke. Indeed, approximately 60% of patients with diagnosis of stroke suffers from hand sensorimotor impairment. In the last years, new approaches in neurorehabilitation field has been permitted to enhance hand motor recovery. Wearable devices permit to apply sensors to the patient's body for monitoring the kinematic and dynamic characteristics of patient's motion. Moreover, wearable sensors combined with electrodes detecting muscle activation (i.e. surface electromyography - sEMG) permit to provide biofeedback to the patient to improve motor recovery.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effect of using REMO® (Morecognition srl, Turin, Italy) device in hand motor rehabilitation.

The device REMO® is an armband composed by 8 bipolar electrodes able to record and process the electromyography of forearm muscles. The patterns of muscle activations are classified and used to perform sEMG-biofeedback exercises in stroke rehabilitation training. The device is developed by clinicians of IRCCS San Camillo Hospital and Morecognition Srl.

A total of 20 patients with first diagnosis of stroke and with no other neurological diagnosis or severe cognitive impairment has been enrolled. The patients are tested with REMO® and if they are able to control at least one movements, they are enrolled in the longitudinal pilot study. The treatment consists in 15 sessions, 1hour/day, for 5 days/week, for 3 weeks. The patients are clinically evaluated before and after the REMO® treatment to define clinical effect of the sEMG-biofeedback training.

ELIGIBILITY:
Inclusion Criteria:

* Single ischemic or haemorrhagic stroke
* able to control at least 1 movement with REMO (i.e. able to cross the pre-defined empirical threshold (10%) of the ratio between the maximum voluntary contraction (MVC) of the movement and the EMG recording during baseline (i.e. rest position)

Exclusion Criteria:

* Untreated epilepsy;
* Major depressive disorder;
* Fractures;
* Traumatic Brain Injury;
* Severe Ideomotor Apraxia;
* Severe Neglect;
* Severe impairment of verbal comprehension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity | Change from baseline, at 3 weeks (15 sessions).
  Fugl-Meyer Upper Extremity is a stroke-specific scale which assesses the upper limb motor functioning in patients with post-stroke hemiplegia. There are 3 values: 0 (severe impairment), 1 (moderate impairment), 2 (preserved function). The minimum value is 0 points, which corresponds to upper limb hemiplegia. The maximum value is 66 points, which corresponds to normal motor performance.

SECONDARY OUTCOMES:
Fugl-Meyer - sensation | Change from baseline, at 3 weeks (15 sessions).
  Sensation of the hemiparetic side is measured by means of the Fugl-Meyer Scale. There are 3 values: 0 (severe impairment), 1 (moderate impairment), 2 (preserved function). The minimum value is 0 points, which corresponds to completely impaired sensory functioning. The maximum value is 24 points, which corresponds to normal sensory functioning.
Fugl-Meyer - pain and Range of Motion | Change from baseline, at 3 weeks (15 sessions).
  Pain and Range of Motion of the hemiparetic upper limb is measured by means of the Fugl-Meyer Scale. There are 3 values: 0 (severe impairment), 1 (moderate impairment), 2 (preserved function). The minimum value is 0 points, which corresponds to maximum level of pain and restriction. The maximum value is 48 points, which corresponds to no pain and normal range of motion.
Box and Blocks Test | Change from baseline, at 3 weeks (15 sessions).
  The patient has to carry as much cubes as possible, one by one, from a container to another one in one minute. The test is performed with both hands.
Reaching Performance Scale | Change from baseline, at 3 weeks (15 sessions).
  Reaching Performance Scale assesses the ability of subjects to reach an object (a cone). The cone is placed at both 4-cm (close) and 30-cm (far) distance from the subject. The subject is asked to reach and grab the cone if possible. The observer evaluates the quality of reaching instead of the grip strength. The minimum value is 0 points, which corresponds to incapacity of any ability of reaching an object. The maximum value is 36 points, which corresponds to the preservation of the ability of reaching an object.
Modified Ashworth Scale | Change from baseline, at 3 weeks (15 sessions).
  Spasticity is measured using the Modified Ashworth Scale of five muscles: Pectoralis major, biceps, wrist flexors, flexor digitorum superficialis, flexor digitorum profundus (Total score = 20 points). The therapist evaluates the spasticity of each muscles. There are 5 values: 0 (no increase in muscle tone), 1 (slight increase in muscle tone), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone), 4 (affected part rigid in flexion or extension).
Nine Hole Pegboard Test | Change from baseline, at 3 weeks (15 sessions).
  Nine Hole Pegboard Test measures the dexterity of the hand. Patient should insert 9 pins in the board. There are 9 pins. The number of pins inserted in 50 sec are registered or if the patient inserted 9 pins, then the time is registered.
Functional Independence Measure | Change from baseline, at 3 weeks (15 sessions).
  Functional Independence Measure scale is an 18-item scale that assesses the degree of independence in carrying out activities of daily living. There are 7 values: 1 (Total Assistance or not Testable), 2 (Maximal Assistance), 3 (Moderate Assistance), 4 (Minimal Assistance), 5 (Supervision), 6 (Modified Independence), 7 (Complete Independence). The minimum values is 18 points, which corresponds to the lower level of independence in activities of daily living. The maximum value is 126 points, which corresponds to the maximum level of independence in activities of daily living.
Number of movements controlled by REMO® device | Change from baseline, at 3 weeks (15 sessions).
  The patient is able to control a movement with the device if he crosses the pre-defined empirical threshold (10%) of the ratio between the maximum voluntary contraction (MVC) of the movement and the sEMG recording during baseline (i.e. rest position).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Turolla, PhD, Principal Investigator — IRCCS San Camillo Hospital
Locations (1):
- IRCCS San Camillo Hospital, Venice-Lido, Venice, Italy

REFERENCES:
- [Background] Celadon N, Dosen S, Binder I, Ariano P, Farina D. Proportional estimation of finger movements from high-density surface electromyography. J Neuroeng Rehabil. 2016 Aug 4;13(1):73. doi: 10.1186/s12984-016-0172-3. PMID 27488270
- [Background] Paleari M, Di Girolamo M, Celadon N, Favetto A, Ariano P. On optimal electrode configuration to estimate hand movements from forearm surface electromyography. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:6086-9. doi: 10.1109/EMBC.2015.7319780. PMID 26737680
- [Background] Di Girolamo M, Celadon N, Appendino S, Turolla A. and Ariano P. EMG-based biofeedback system for motor rehabilitation: A pilot study,. IEEE Biomedical Circuits and Systems Conference (BioCAS). 2017; pp. 1-4, doi: 10.1109/BIOCAS.2017.8325086.
- [Background] Parker J, Powell L, Mawson S. Effectiveness of Upper Limb Wearable Technology for Improving Activity and Participation in Adult Stroke Survivors: Systematic Review. J Med Internet Res. 2020 Jan 8;22(1):e15981. doi: 10.2196/15981. PMID 31913131
- [Background] Maceira-Elvira P, Popa T, Schmid AC, Hummel FC. Wearable technology in stroke rehabilitation: towards improved diagnosis and treatment of upper-limb motor impairment. J Neuroeng Rehabil. 2019 Nov 19;16(1):142. doi: 10.1186/s12984-019-0612-y. PMID 31744553